CLINICAL TRIAL: NCT03222908
Title: Evaluation of Surgical Outcomes in Patients Undergoing Pre-commitment and Social Contracting for Smoking Cessation
Brief Title: Perioperative Smoking Cessation Interventions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment and lack of interest
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00076125
Record Dates: First submitted 2017-07-18; First posted 2017-07-19 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Smoking Cessation; Perioperative/Postoperative Complications
Keywords: Behavior; Perioperative/Postoperative Complications; contract agreement; implementation intentions; precommitment; smoking cessation
MeSH Terms: conditions — Smoking Cessation; Postoperative Complications; Behavior

STUDY DESIGN:
Intervention Model Description: randomized control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control: Prescriptive Advice (No Intervention): Amenable patients will be enrolled into the study, their intervention will be current standard of care smoking cessation counseling by their surgeon, they will undergo 3 urine tests and a chart review for outcomes.
- Intervention1: Contract Agreement (Experimental): Amenable patients will be enrolled into the study, their intervention will be a smoking cessation contract with their surgeon, they will undergo 3 urine tests and a chart review for outcomes.
  Interventions: Behavioral: Intervention1: Contract Agreement
- Intervention2: Implementation Intentions (Experimental): Amenable patients will be enrolled into the study, their intervention will be a worksheet to fill out with their smoking cessation implementation intentions that will be signed by patient and surgeon, they will undergo 3 urine tests and a chart review for outcomes.
  Interventions: Behavioral: Intervention2: Implementation Intentions

INTERVENTIONS:
Behavioral: Intervention1: Contract Agreement — Smoking Cessation Contract
  Arms: Intervention1: Contract Agreement
Behavioral: Intervention2: Implementation Intentions — Smoking Cessation Contract with worksheet for implementation intentions
  Arms: Intervention2: Implementation Intentions

SUMMARY:
To assess impact of behavioral economic principles of precommitment, implementation intentions, and social contracting on smoking cessation for patients undergoing surgery.

DETAILED DESCRIPTION:
Purpose & Objective: Behavioral interventions in surgical patients are an opportunity to improve outcomes through decreased complications, with measurable economic impact. Smoking cessation is one of the most desirable long-term health behaviors for adults with potential substantial impact on postoperative complications

Study Activity & Population Group: The investigators propose a precommitment contractual agreement implementing behavioral economic principles at the preoperative appointment for active tobacco users undergoing an operation and assessing for ability to quit smoking with testing on the day of surgery, and the durability of cessation over the postoperative course as measured with urine nicotine testing at follow up appointments. The population of interest is adults who currently smoke tobacco or vaporized nicotine who are scheduled to undergo a major operation. The control group is standard of care; prescriptive advice to quit smoking. The intervention is contract agreement for preoperative cessation.

Data Analysis & Risk Issues: Following informed consent patients will be randomized to control or intervention groups, baseline urine nicotine tests will be performed in clinic. Urine nicotine testing will be performed on the day of enrollment, the day of their operation, and at their one-month follow up appointments. Thirty-day outcomes will be evaluated by retrospective chart review.

ELIGIBILITY:
Inclusion Criteria:

* active tobacco use
* preoperative appointment for an operation within 6 weeks

Exclusion Criteria:

* active enrollment in tobacco cessation program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Smoking Cessation | day of surgery
  Smoking Cessation on Day of Surgery: quantitative point of care urine cotinine test
Smoking Cessation | day of first postoperative appointment
  Smoking Cessation on first postoperative follow up appointment: quantitative point of care urine cotinine test

SECONDARY OUTCOMES:
Postoperative Complications | 30 days postoperatively
  National Surgical Quality Improvement Project postoperative complications: based on patient chart review

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R Mantyh, MD, Principal Investigator — DUKE DEPARTMENT OF SURGERY
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
no plan to share data